CLINICAL TRIAL: NCT01070511
Title: Functional Muscle Ischemia and PDE5A Inhibition in Becker Muscular Dystrophy
Brief Title: Tadalafil in Becker Muscular Dystrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Principal Investigator, Ron Victor, Director Hypertension Center, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MDA 158944; NCT02207283 (obsolete NCT alias); NCT03076814 (obsolete NCT alias)
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Becker Muscular Dystrophy
Keywords: Muscular Dystrophy; Tadalafil
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Experimental)
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tadalafil will be administered orally on two consecutive days. The first dose-10 mg- will be administered the afternoon before the study. The second dose -20 mg-will be administered the morning of the study.
  Other Names: Cialis
  Arms: Tadalafil
Drug: Placebo — A placebo pill will be administered orally on two consecutive days. The first pill will be administered the afternoon before the study. The second pill will be administered the morning of the study.
  Arms: Placebo

SUMMARY:
Summary for Patients: This study, funded by the Muscular Dystrophy Association, is intended to build on recent findings published in the journal Nature showing beneficial effects of tadalafil (also known as Cialis) in mice with an animal version of Duchenne and Becker muscular dystrophies. Only two doses of tadalafil improved muscle blood flow, allowing the dystrophic mice to perform more exercise with less muscle injury. This new short-term clinical trial will move the testing from animals to human patients with Becker muscular dystrophy and examine the effects of acute tadalafil dosing on muscle blood flow during a bout of exercise. Patients will take two doses of tadalafil prior to exercising. Then doctors will measure whether muscles receive increased blood flow and therefore are better protected during exercise.

Scientific Hypothesis: In patients with Becker muscular dystrophy (particularly those with dystrophin gene mutations between exons 41-46), loss of sarcolemmal nitric oxide synthase engenders functional muscle ischemia and thus muscle edema after an acute bout of exercise. The investigators further hypothesize that PDE5A inhibition, which boosts nitric oxide-cGMP signaling, constitutes an effective new countermeasure for these patients.

DETAILED DESCRIPTION:
There are 2 phases to this research project: (1) an initial baseline study to compare patients with Becker muscular dystrophy against healthy control subjects, and (2) a subsequent brief treatment trial only in the muscular dystrophy patients (healthy controls will not participate in this second phase of the study).

The baseline study involves an intake history, physical examination, and phlebotomy for blood chemistries and DNA followed by (a) MRI scans of the forearm muscles before and after a brief bout of handgrip exercise approximately 1-1.5 hours to complete), and (b) non-invasive forearm blood flow studies (Near Infrared Spectroscopy, Doppler Ultrasound) before and after a brief bout of handgrip exercise (approximately 3-5 hours to complete). Blood flow studies will be performed with the subject's lower body enclosed in an airtight chamber. Blood flow and oxygen delivery to the forearm muscles will be measured before and during application of lower body negative pressure at rest and during handgrip exercise. Lower body negative pressure simulates the blood flow changes that normally occur when a person sits up after lying down.

The results of the baseline study will determine which patients meet preset eligibility criteria to participate in the medication phase of the study. These criteria include (1) normal kidney and liver function tests and normal BNP levels (the latter to exclude heart failure), and (2) abnormal MRI and blood flow responses to handgrip exercise. Eligible patients will be asked to repeat the above laboratory procedures on two more study days: one day after receiving 2 pills of tadalafil (a PDE5A inhibitor that is longer-lasting than Viagra) and another day after receiving 2 placebo pills. Study procedures can be broken up into two separate days for scheduling purposes and/or to avoid fatigue. Patients completing the trial will receive both study medications and the order will be random.

In summary, healthy control subjects will only undergo the baseline study whereas Becker muscular dystrophy patients completing all phases of the project will have 3 separate study days (baseline, tadalafil, and placebo) and 2 medication visits (to receive the study medication and have their blood pressure checked by a study physician). Study days will be separated by at least two weeks to allow time for test results, to rest the forearm muscles between exercise bouts, and to ensure complete elimination of tadalafil.

We plan to enroll 24 adult men with Becker muscular dystrophy, of whom 12 men will have dystrophin gene deletions between exons 41-46, and 24 healthy control subjects.

ELIGIBILITY:
Becker Muscular Dystrophy Patients

* Men 18-55 years of age with a pre-existing diagnosis of Becker Muscular Dystrophy by a clinical neurologist (based on clinical criteria plus previous muscle biopsy analysis and/or DNA analysis).

Healthy Controls

* Men 18-55 years of age with no known medical conditions

Criteria for exclusion of subjects (both patients and controls)

* Any evidence of cardiopulmonary disease by history or by physical examination
* History of hypertension or blood pressure averaging ≥140/90 mmHg
* Diabetes mellitus or other systemic illness
* Heart failure by clinical exam, elevated BNP, or heart failure medication
* Serum creatinine ≥ 1.5 mg/dL
* Any history of substance abuse (including alcohol)
* Any history of psychiatric illness
* Contraindications to tadalafil (use of nitrates, alpha-blockers, other PDE5A inhibitors, or potent inhibitors of CYP3A4 such as ketoconazole or ritonavir)
* Contraindications to MRI (claustrophobia, metal implants, or seizure disorder)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reflex decrease in muscle tissue oxygenation (i.e., adrenergic vasoconstriction) during rhythmic handgrip exercise measured by Near Infrared Spectroscopy (NIR). | measured at a minimum of 2 week intervals for a minimum of 6 weeks total (for subjects with BMD)

SECONDARY OUTCOMES:
Change in forearm muscle water content by magnetic resonance imaging (MRI). | measured at a minimum of 2 week intervals for a minimum of 6 weeks total (for subjects with BMD)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California